CLINICAL TRIAL: NCT07289516
Title: The Effect Of Music Played To Women Who Gave Birth By Cesarean Section On Pain, Comfort And Mother İnfant Bonding Level İn The Early Period
Brief Title: Effect Of Lıstenıng to Musıc on Women Gıvıng Bırth By Cesarean Sectıon: Paın, Comfort And Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ebru Unal, Expert Midwife, Principal Investigator, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BU-SBE-EU-001
Record Dates: First submitted 2025-01-29; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Delivery; Music Listening
Keywords: pain; bonding; comfort; music; cesarean delivery; midwifery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Women in the experimental group listened to music for 20 minutes twice, at the 8th and 16th postpartum hours. Women in the control group received routine midwifery/nursing care practices provided in the clinic after cesarean delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, women were exposed to music for 20 minutes twice, at the 8th and 16th hours postpartum. At the 8th postpartum hour, the Personal Information Form, Visual Analog Scale, Postpartum Comfort Scale, and Maternal-Infant Attachment Scale were administered. Music was played for 20 minutes, and routine midwifery care was provided. Thirty minutes after the intervention, the Visual Analog Scale was administered again. At the 16th postpartum hour, the Visual Analog Scale, routine midwifery care, and another 20-minute music session were conducted. Thirty minutes after this session, the Visual Analog Scale, Postpartum Comfort Scale, and Maternal-Infant Attachment Scale were applied.
  Interventions: Behavioral: Music intervention
- Control Group (No Intervention): In the control group, at the 8th postpartum hour, the Personal Information Form, Visual Analog Scale, Postpartum Comfort Scale, and Maternal-Infant Attachment Scale were administered. Routine midwifery care was provided. Thirty minutes after the intervention, the Visual Analog Scale was applied again. At the 16th postpartum hour, the Visual Analog Scale and routine midwifery care were administered. Thirty minutes after this intervention, the Visual Analog Scale, Postpartum Comfort Scale, and Maternal-Infant Attachment Scale were administered.

INTERVENTIONS:
Behavioral: Music intervention — To play music
  Arms: Experimental Group

SUMMARY:
This study aims to evaluate the effect of music played for women who undergo cesarean delivery on their early-stage pain, comfort, and mother-infant bonding levels. The study was conducted with 62 women who had cesarean deliveries and were hospitalized in the Obstetrics Unit of Bilecik Training and Research Hospital. Participants were randomly assigned to either an experimental group or a control group. Music in the Acemaşiran mode was played for 20 minutes twice, at the 8th and 16th postpartum hours for the experimental group, while the control group received routine midwifery/nursing care practices provided in the clinic after cesarean delivery. The study is designed to assess whether listening to music after cesarean delivery influences postoperative pain, comfort, and mother-infant bonding levels.

DETAILED DESCRIPTION:
This study is designed to evaluate the effect of music played for women undergoing cesarean section on early-stage pain, comfort, and mother-infant bonding. The study included a total of 62 women who had cesarean deliveries and were admitted to the Obstetrics and Gynecology Department of Bilecik Training and Research Hospital. Participants were randomly assigned to an experimental group (n=31) and a control group (n=31).

Data are collected using the Descriptive Information Form, Visual Analog Scale (VAS), Postpartum Comfort Scale (PPCS), and Mother-Infant Attachment Scale (MBIS). The data will be analyzed using IBM SPSS V23 and JAMOVI V2.3.21 software.

The study is designed to compare the effects of listening to music in the Acemaşiran mode with standard postpartum care after cesarean delivery. The intervention involves listening to music for 20 minutes at the 8th and 16th postpartum hours in the experimental group, while the control group receives routine midwifery/nursing care practices.

The following hypotheses will be tested:

H1-a: Listening to music affects the pain levels of women after cesarean delivery.

H1-b: Listening to music affects the comfort levels of women after cesarean delivery.

H1-c: Listening to music affects the physical comfort levels of women after cesarean delivery.

H1-d: Listening to music affects the sociocultural comfort levels of women after cesarean delivery.

H1-e: Listening to music affects the psychospiritual comfort levels of women after cesarean delivery.

H1-f: Listening to music affects the mother-infant bonding relationship of women after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participants,
* Undergoing cesarean delivery between 38-40 weeks of gestation,
* Aged between 18-45 years,
* Literate and fluent in Turkish,
* Experiencing no complications during or after the cesarean procedure,
* Having an uncomplicated pregnancy,
* Free of chronic illnesses,
* Without any auditory or visual impairments,
* Without a diagnosed mental health condition,
* Giving birth to a single, healthy, and live newborn.

Exclusion Criteria:

* Individuals who do not consent to participate,
* Those with any cognitive, sensory, or verbal impairments that hinder communication,
* Diagnosed with any medical condition during pregnancy,
* Experiencing postpartum complications affecting either the mother or the fetus,
* Having a newborn admitted to the neonatal intensive care unit,
* Experiencing chronic pain,
* Individuals with hearing impairments,
* Diagnosed with psychiatric or chronic illnesses.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by the Visual Analog Scale (VAS) | Baseline (before intervention), 30 minutes after the first music session, and 30 minutes after the second music session.
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10-point scale ranging from 0 (no pain) to 10 (worst possible pain). Higher scores indicate greater pain intensity.
Change in Postpartum Comfort Level Measured by the Postpartum Comfort Scale (PPCS) | 8th and 16th postpartum hours.
  The Postpartum Comfort Scale (PPCS) is a 34-item Likert-type scale that assesses overall comfort levels of postpartum women. Each item is scored between 1 (disagree) and 4 (strongly agree), with total scores ranging from 34 to 136. Higher scores indicate higher comfort levels.
Change in Mother-Infant Bonding Measured by the Mother-Infant Bonding Scale (MIBS) | 16th postpartum hour.
  The Mother-Infant Bonding Scale (MIBS) is an 8-item scale measuring maternal emotional bonding toward the infant. Each item is scored from 0 to 3, with total scores ranging from 0 to 24. Higher scores indicate weaker bonding (worse outcome).

SECONDARY OUTCOMES:
Change in Physical Comfort Level Measured by the Physical Comfort Subscale of the Postpartum Comfort Scale (PPCS) | 8th and 16th postpartum hours.
  The Physical Comfort Subscale of the Postpartum Comfort Scale (PPCS) assesses physical well-being and recovery in postpartum women. Items are scored from 1 (disagree) to 4 (strongly agree), and total scores range from 10 to 40. Higher scores indicate greater physical comfort.
Change in Sociocultural Comfort Level Measured by the Sociocultural Comfort Subscale of the Postpartum Comfort Scale (PPCS) | 8th and 16th postpartum hours.
  The Sociocultural Comfort Subscale of the Postpartum Comfort Scale (PPCS) evaluates the sociocultural adaptation and support experienced by postpartum women. Each item is scored from 1 to 4, and total scores range from 8 to 32. Higher scores indicate greater sociocultural comfort.
Change in Psychospiritual Comfort Level Measured by the Psychospiritual Comfort Subscale of the Postpartum Comfort Scale (PPCS) | 8th and 16th postpartum hours.
  The Psychospiritual Comfort Subscale of the Postpartum Comfort Scale (PPCS) assesses emotional, spiritual, and psychological comfort in postpartum women. Each item is scored from 1 to 4, with total scores ranging from 10 to 40. Higher scores indicate greater psychospiritual comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin PALAS KARACA, Associate Professor, Principal Investigator — Balikesir University
Locations (1):
- Bilecik Training and Research Hospital, Bilecik, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No